CLINICAL TRIAL: NCT03599362
Title: Nivolumab, Cabiralizumab, and Stereotactic Body Radiotherapy (SBRT) for Locally Advanced Unresectable Pancreatic Cancer
Brief Title: Study of Nivolumab, Cabiralizumab, and Stereotactic Body Radiotherapy (SBRT) for Locally Advanced Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI departure from institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-01430
Record Dates: First submitted 2018-07-10; First posted 2018-07-26 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; cabiralizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi Agent Chemotherapy Cancer Patients (Experimental): Subjects will be enrolled into this study following completion of 2-6 months of multi agent chemotherapy with documentation of stable or responsive disease.
  Interventions: Drug: Nivolumab + Cabiralizumab; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Nivolumab + Cabiralizumab — Will be administered on Day 1 and Day 14; Subjects will continue treatment every 2 weeks with subsequent imaging every 8 weeks.
Radiation: Stereotactic Body Radiotherapy (SBRT) — Patients will be simulated supine with the addition of a 4D C T if appropriate. A stereotactic immobilization device with abdominal compression will be used.

SUMMARY:
A multi-institutional, single arm phase II study of nivolumab, cabiralizumab and stereotactic body radiotherapy (SBRT) in patients with LAUPC. The purpose of this study is to determine the safety and tolerability of combined cabiralizumab, nivolumab and radiotherapy in the treatment of locally advanced pancreatic cancer. Investigators will also estimate the surgical resection rate following treatment with combined cabiralizumab, nivolumab and radiotherapy in subjects with locally advanced unresectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced, unresectable pancreatic cancer as defined by NCCN Guidelines 3.2017
* Locally advanced unresectable disease is defined by the NCCN as:
* Tumors of the head that have greater than 180 degrees of SMA encasement or any celiac abutment, unreconstructable SMV or portal occlusion, or aortic invasion or encasement.
* Tumors of the body with SMA or celiac encasement of greater than 180 degrees, unreconstructable SMV or portal occlusion, or aortic invasion.
* Tumors of the tail with SMA or celiac encasement of greater than 180 degrees. Irrespective of location, all tumors with evidence of nodal metastasis outside of the resection field are deemed unresectable.
* Patients must agree to pretreatment and on treatment tumor biopsy
* ECOG performance status of 0 or 1
* Completion of at least 2 months, but no more than 6 months of standard induction chemotherapy for LAPC, which must include either FOLFIRINOX or gemcitabine and nab- paclitaxel, preferably within 2-4 weeks but no longer than 8 weeks.
* Normal organ and marrow function as defined below:
* absolute neutrophil count ≥ 1,500/mm3
* platelets ≥ 100,000/mm3
* total bilirubin ≤ 1.5 x institutional upper limit of normal (except participants with Gilbert's syndrome who must have normal direct bilirubin)
* AST(SGOT) and ALT(SGPT) ≤ 2 × institutional upper limit of normal
* creatinine ≤ 1.5 mg/ dL OR
* creatinine clearance≥ 30 mL/min (as estimated by Cockcroft Gault Equation)
* Ability to understand and sign a written informed consent document. Participant must have willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Women of childbrearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) and for a total of 5 months post-treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (see appendix 1) for the duration of treatment with study treatment(s) and for a total of 7 months posttreatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Resectable, borderline resectable or metastatic disease
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease.

Note: Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted.

* Current or history of clinically significant muscle disorders (eg, myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:
* Myocardial infarction or stroke/transient ischemic attack within the past 6 months
* Uncontrolled angina within the past 3 months
* Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
* Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
* Evidence of uncontrolled, active infection, requiring parenteral anti-bacterial, anti-viral or anti-fungal therapy ≤ 7 days prior to administration of study medication.
* Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis.
* Participants with active, known, or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussing with the Principal Investigator.
* Concomitant use of statins while on study. However, a patient using statins for over 3 months prior to study drug administration and in stable status without CK rise may be permitted to enroll.
* Non-oncology vaccine therapies for prevention of infectious diseases (eg, human papillomay virus vaccine) within 4 weeks of study drug administration. The inactivated seasonal influenza vaccine can be given to patients before treatment and while on therapy without restriction. Influenza vaccines containing live virus or other clinically indicated vaccinations for infectious diseases (ie, pneumovax, varicella, etc) may be permitted, but must be discussed with the principal investigator and may require a study drug washout period prior to and after administration of vaccine.
* Known human immunodeficiency virus (HIV), known active hepatitis A, or known hepatitis B or C infection.
* History of acute diverticulitis within the last 6 months, or current chronic diarrhea
* Pregnant or lactating women.
* Women of childbearing potential (WOCBP) with either a positive or no pregnancy test (serum or urine) at baseline. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.)
* WOCBP who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy (see appendix 1) for the entire study period and for at least 5 months after the last dose of investigational product. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but still must undergo pregnancy testing as described in section - Sexually active fertile men not using effective birth control if their partners are WOCBP
* History of primary immunodeficiency.
* History of organ allograft or allogeneic bone marrow transplant.
* Any prior radiation therapy, immunotherapy, or biologic ('targeted') therapy for treatment of the patient's pancreatic tumor. Patient should have received either FOLFIRINOX or gemcitabine and nab-paclitaxel prior to enrollment.
* Treatment for other invasive carcinomas within the last five years who are at greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.
* History of allergy to study treatments or any of its components
* Known history of sensitivity to infusions containing Tween 20 (polysorbate 20) and Tween 80 (polysorbate 80)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multi Agent Chemotherapy Cancer Patients
Started | 7
Completed | 4
Not Completed | 3
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Multi Agent Chemotherapy Cancer Patients
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 68 [37 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Unacceptable Toxicity
Description: Measure of safety of combined cabiralizumab, nivolumab and radiotherapy in the treatment of locally advanced pancreatic cancer measured by unacceptable toxicity, which includes:
  * Grade 3 fatigue lasting > 2 Weeks
  * Grade 3 Nausea lasting > 7 days despite maximal medical management
  * Grade 3 or more anorexia
  * Grade 3 or more vomiting
  * Grade 3 or more diarrhea
  * Grade 3 or more pancreatitis
  * Grade 3 abdominal pain
  * Grade 3 or more radiation dermatitis
  * Grade 3 or more GI hemorrhage
  * Grade 3 or more GI fistula
  * Grade 3 or more GI stenosis
  * Grade 3 or more GI perforation
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Multi Agent Chemotherapy Cancer Patients
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Participants Who Proceeded to Surgical Resection
Description: Surgical resection rate following treatment with combined cabiralizumab, nivolumab and radiotherapy in subjects with locally advanced unresectable pancreatic cancer.
  This will be measured by tabulating adverse events
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Multi Agent Chemotherapy Cancer Patients
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Multi Agent Chemotherapy Cancer Patients
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multi Agent Chemotherapy Cancer Patients (N=4)
Liver dysfunction (Hepatobiliary disorders) | 1
Chest Pain (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Multi Agent Chemotherapy Cancer Patients (N=4)
Abdominal Pain (Gastrointestinal disorders) | 2
Agitation (Psychiatric disorders) | 1
Increase in ALT (Investigations) | 4
Increase in AST (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Increase in Alkaline Phosphatase (Investigations) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Chills (General disorders) | 2
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Increase in CPK (Investigations) | 4
Increase in Creatinine (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ear and Labyrinth Disorder (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Edema Face (General disorders) | 1
Epis Taxis (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 1
Gait Disturbance (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
General Disorders and Administration Site Conditions (General disorders) | 1
Headache (Nervous system disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Investigations) | 1
Hyponatremia (Investigations) | 1
Increase in Lipase (Investigations) | 4
Localized Edema (General disorders) | 1
Decrease in Lymphocyte Count (Investigations) | 3
Nausea (Gastrointestinal disorders) | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Periorbital Edema (Eye disorders) | 1
Decrease in Platelet Count (Investigations) | 2
Pruritus (General disorders) | 1
Rash Maculo (Skin and subcutaneous tissue disorders) | 2
Increase in Serum Amylase (Investigations) | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Decrease in WBC (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03599362/Prot_SAP_000.pdf